CLINICAL TRIAL: NCT04058535
Title: A Phase I Clinical Study of ALT-L9 in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Clinical Study of ALT-L9 to Determine Safety, Efficacy and Pharmacokinetics in Neovascular AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alteogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-L9-01
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALT-L9 (Experimental): Intravitreal injection of ALT-L9 50 ul, every 4 weeks
  Interventions: Biological: ALT-L9
- Eylea (Active Comparator): Intravitreal injection of Eylea 50 ul, every 4 weeks
  Interventions: Biological: Eylea

INTERVENTIONS:
Biological: Eylea — Aflibercept
  Arms: Eylea
Biological: ALT-L9 — Aflibercept biosimilar
  Arms: ALT-L9

SUMMARY:
To evaluate the safety, efficacy and pharmacokinetics of repeated intravitreal administration of ALT-L9 2 mg/50uL compared with Eylea in patients with neovascular Age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50years old or more at the time of consent.
2. Patients with any history of anti-VEGF treatment(Aflibercept, Bevacizumab, Ranibizumab) for neovascular AMD in the study eye.
3. Patients who were treated with the last anti-VEGF at least 8 weeks prior to study drug administration.
4. Patients with untreated active primary subfoveal CNV lesions secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by FA, ICGA, and/or SD-OCT in the study eye at the start of the screening visit.
5. Patients with subretinal, intraretinal, or subretinal pigment epithelium fluid as assessed by SD-OCT in the study eye at the start of the screening visit.
6. Patients with ETDRS best-corrected visual acuity of 20/40 to 20/320 (letter score of 73 to 25) in the study eye at the start of the administration of the study drug.
7. Patients with ETDRS best-corrected visual acuity of 20/400 (letter score 20) or better in the fellow eye at the start of the administration of the study drug.
8. Patients who provide written informed consent to participate in this clinical study

Exclusion Criteria:

1. Patients who have received any prior ocular (in the study eye) or systemic treatment for neovascular AMD within 8 weeks from the baseline date except dietary supplements or vitamins.
2. Patients who have received any surgery for neovascular AMD.
3. Patients with any current or history of macular or retinal disease other than neovascular AMD (eg, diabetic macular edema, retinal vein occlusion, pathological myopia, angioid streaks, ocular histoplasmosis, trauma, retinal detachment, epiretinal membrane, macular hole, central serous chorioretinopathy, Choroidal rupture, Multiple network choroiditis, proliferative diabetic retinopathy) in the study eye.
4. Patients with scar, fibrosis, or atrophy involving the center of the fovea in the study eye that might interfere with visual acuity.
5. Patients with hemorrhage under the fovea or subretinal hemorrhage 50% or more of the total lesion area in the study eye.
6. Patients with retinal pigment epithelial tears or rips involving the macula in the study eye.
7. Patients with a history of any vitreous hemorrhage or rhegmatogenous retinal detachment in the study eye within 4 weeks before the start of the administration of the study drug.
8. Patients who have received panretinal photocoagulation in the study eye.
9. Patients who have received vitreous surgery in the study eye.
10. Patients with a history of corneal transplant or corneal dystrophy in the study eye.
11. Patients who have received cataract surgery or Lasik in the study eye within 90 days before the start of the administration of the study drug.
12. Patients who have received trabeculectomy or other filtration surgery in the study eye
13. Patients with poorly controlled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye.
14. Patients with significant media opacities, including cataract, in the study eye that might interfere with visual acuity, assessment of safety, or fundus photography considered by the principal investigator or investigator.
15. Patients with any diseases in the study eye that could have compromised visual acuity such as amblyopia and anterior ischemic optic neuropathy considered by the principal investigator or investigator.
16. Patients with cataract in the study eye that could have required medical or surgical intervention during the course of the study considered by the principal investigator or investigator.
17. Patients with aphakia with absence of posterior capsule in the study eye.
18. Patients who have received therapeutic radiation in the region of the study eye.
19. Patients who use topical ocular corticosteroids for 30, or more, consecutive days within 90 days before the screening visit, or have a plan or actual use for 30 or more consecutive days during the course of the study in the study eye.

    Criteria for fellow eye or either eye:
20. Patients with any active intraocular or periocular infection or intraocular inflammation in either eye (eg, infectious blepharitis, infectious conjunctivitis, keratitis, scleritis, endophthalmitis).
21. Patients with a history of uveitis in either eye.
22. Patients with a concurrent or history of scleromalacia in either eye.
23. Patients who have received anti-VEGF medication in the fellow eye within 8 weeks before the start of the administration of the study drug.

    Other criteria:
24. Patients who use systemic corticosteroids for 30 or more consecutive days within 90 days before the Screening Visit, or have a plan or actual use for 30 or more consecutive days during the course of the study. Inhaled steroids were permitted.
25. Patients who use steroid(except systemic or inhaled steroid) within 6 months, or have a plan for use of steroid during the course of the study.
26. Patients with poorly controlled hypertension. (defined as systolic BP is 160 mmHg or more or diastolic BP is 100 mmHg or more despite medication)
27. Patients with a serious liver, kidney or cardiovascular disorders considered by the principal investigator or investigator.
28. Patients with a concurrent or history of malignancy within 5 years before informed consent.
29. Patients with drug abuse (defined as use of illegal drugs) or alcohol dependence or a history of these conditions.
30. Patients with a history of clinically significant drug hypersensitivity.
31. Patients with a history of allergy to aflibercept, fluorescein, indocyanine green and povidone iodine.
32. Patients with any contraindications described in aflibercept package insert.
33. Females who are pregnant, breastfeeding, or of childbearing potential, unwilling to practice adequate contraception throughout the study.
34. Patients with type 1 diabetes or increase of HbA1c(>12%).
35. Patients who have received any other investigational drug within 12 weeks before screening visit.
36. Other patients considered by the principal investigator or investigator to be inappropriate as subjects.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Occurrences of adverse events | 8 weeks
  Check the adverse events in study eye at the assessment points after triple administration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea